CLINICAL TRIAL: NCT04792294
Title: Multicenter Analysis of Efficacy and Outcomes of Extracorporeal Photopheresis as Treatment of Chronic Lung Allograft Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alberto Benazzo, MD, Principal Investigator, Medical University of Vienna
Other Study IDs: 1541/2020
Record Dates: First submitted 2021-02-25; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Lung Transplant Rejection
MeSH Terms: interventions — Photopheresis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Lung transplant recipients with chronic lung allograft dysfunction: Lung transplant recipients with chronic lung allograft dysfunction, who underwent extracorporeal photopheresis
  Interventions: Device: Extracorporeal photopheresis

INTERVENTIONS:
Device: Extracorporeal photopheresis — ECP can be used as second-line treatment in patients unresponsive to azithromycin. ECP has been firstly developed for treatment of cutaneous T cell lymphomas and later used in a variety of other indications including solid organ transplantation. The process starts with leukapheresis, followed by incubation of the isolated cells with 8-methoxypsoralen (8-MOP) and subsequent activation of 8-MOP with ultraviolet A radiation. At the end, the cells are reinfused into the patient. 8-MOP is a biologically inert substance, but in the presence of UVA light it cross-links DNA by forming covalent bonds with pyrimidine bases and causes apoptosis.

SUMMARY:
Lung transplantation is an established therapy for end-stage lung disease such as chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, cystic fibrosis and pulmonary hypertension. However, Chronic Lung Allograft Dysfunction (CLAD) is a major cause of morbidity and mortality in long-term survivors. The 5-year survival rate is reported to be 50%, which is considerably inferior compared to other solid organ transplantation. In addition, the financial burden of CLAD (around 80.000 euro/year for a patient with CLAD) is considerable. No curative therapy is available yet. To date, the two most effective treatment are azithromycin and extracorporeal photopheresis. Azithromycin is used as first-line treatment and it is effective in stopping FEV1 decline, however its effects are only limited to a set of patients. ECP can be used as second-line treatment in patients unresponsive to azithromycin. ECP has been firstly developed for treatment of cutaneous T cell lymphomas and later used in a variety of other indications including solid organ transplantation. The process starts with leukapheresis, followed by incubation of the isolated cells with 8-methoxypsoralen (8-MOP) and subsequent activation of 8-MOP with ultraviolet A radiation. At the end, the cells are reinfused into the patient. 8-MOP is a biologically inert substance, but in the presence of UVA light it cross-links DNA by forming covalent bonds with pyrimidine bases and causes apoptosis. ECP is effective in the palliative treatment of cutaneous T-cell lymphoma but its effectiveness was also shown in several other T-cell-mediated diseases, particularly in the treatment and prevention of acute and chronic graft-versus-host disease. In depth knowledge on the mechanisms whereby ECP manipulates the immune system are still unclear. Most of the experimental studies have been performed in murine models of GvHD. Apoptotic cells isolated during ECP treatment have the potential to induce IL-10 secretion, reduce dendritic cells activation and increase percentage of Tregs. In addition, ECP reduces the production of IL-6 and TNF-α and increases TGF-β production. In lung transplantation, ECP treatment is used as second-line treatment of CLAD and it has the potential to stabilize lung function decline and to improve long-term graft. According to the published literature, however, approximately 30 to 40% of treated recipients did not profit from ECP. Greer and colleagues found that RAS patients as well as rapid lung function decliners showed lower rate of response and worse long-term outcomes. On the contrary in a more recent analysis only BOS diagnosis was associated with better outcomes. A single prospective interventional study was published by our group and it confirmed results from other previous retrospective analysis. Up to now, no clear predictors for response have been identified yet.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of CLAD Adult transplant recipients (>18 years)

Exclusion Criteria:

ECP for other diagnosis Recipients of multi-organ transplantation Recipients of single lung transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant recipients with chronic lung allograft dysfunction who received extracorporeal photopheresis as treatment
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in forced expiratory value in 1 second at 3 months after start of extracorporeal photopheresis | 3 months
  Percentage change in FEV1 within 3 months after start of extracorporeal photopheresis

SECONDARY OUTCOMES:
change in maximal expiratory flow (50%) at 3 months after start of extracorporeal photopheresis | 3 months
  Percentage change in MEF50 within 3 months after start of extracorporeal photopheresis
Change in forced expiratory value in 1 second/dorced vital capacity ratio at 3 months after start of extracorporeal photopheresis | 3 months
  Percentage change in FEV1/FVC within 3 months after start of extracorporeal photopheresis
Change in total lung capacity at 3 months after start of extracorporeal photopheresis | 3 months
  Percentage change in TLC within 3 months after start of extracorporeal photopheresis
Patients' survival | Within 5 years from start of extracorporeal photopheresis
  Patients' survival
Graft survival | Within 5 years from start of extracorporeal photopheresis
  Graft survival
Adverse events on extracorporeal photopheresis | Within 5 years from start of extracorporeal photopheresis
  Adverse events on extracorporeal photopheresis